CLINICAL TRIAL: NCT06900660
Title: Evaluation of the Skin-Beautifying Effects of Collagen Drinks
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Simply Plus Co., Ltd. (Industry)
Collaborators: Chia Nan University of Pharmacy ＆ Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-007-B
Record Dates: First submitted 2025-03-26; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Collagen Drinks (Experimental): The Collagen Drinks contain collagen peptides and antioxidants
  Interventions: Dietary Supplement: Collagen Drinks

INTERVENTIONS:
Dietary Supplement: Collagen Drinks — Dosage: 50 mL/day; duration: 8 weeks

SUMMARY:
This study aims to investigate the skin beauty benefits of collagen drinks in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Healthy people

Exclusion Criteria:

1. Non-volunteer
2. Pregnant and lactating women
3. Hypersensitivity to the assigned product
4. Diagnosed with skin diseases, liver diseases, kinedy disease, and other severe diseases
5. Cosmetic, drug, or food allergies
6. Concurrent aesthetic treatments (e.g., intense pulse light, medical peelings, or laser therapy)
7. Aceepted aesthetic treatments one month ago before the study
8. Chronic sun exposure (over 3 hours/day)
9. The members of the research team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of skin hydration | Week 0, 4, 8
  Corneometer CM825 is used to measure the moisture of upper cheek
Measurement of skin elasticity | Week 0, 4, 8
  Cutometer® is used to measure the skin elasticity of upper cheek
Measurement of skin wrinkles | Week 0, 4, 8
  Visia® skin analysis system is used to measure the skin wrinkles of full face
Measurement of skin pores | Week 0, 4, 8
  Visia® skin analysis system is used to measure the skin spots of full face
Measurement of collagen content | Week 0, 4, 8
  DermaLab® Series SkinLab Combo (Cortex) is employed to measure skin collagen content of upper cheek
Measurement of wrinkles around the eyes | Week 0, 4, 8
  Visia® skin analysis system is used to measure the skin wrinkles around the eyes
Measurement of skin brightness | Week 0, 4, 8
  Chroma Meter MM500 is employed to measure the brightness of upper cheek
Measurement of collagen levels in the blood | Week 0, 8
  Analysis of changes in beauty-related biomarkers in the blood
Measurement of hyaluronic acid levels in the blood | Week 0, 8
  Analysis of changes in beauty-related biomarkers in the blood
Measurement of superoxide dismutase (SOD) levels in the blood | Week 0, 8
  Analysis of changes in beauty-related biomarkers in the blood

SECONDARY OUTCOMES:
The change of self-assessment skin condition | Week 0, 4, 8
  A self-assessment questionnaire was collected and evaluate skin condition

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Principal Investigator — Department of Cosmetic Science, Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No